CLINICAL TRIAL: NCT00848627
Title: Screening for Bladder Cancer
Status: Completed | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Collaborators: M.D. Anderson Cancer Center (Other); University of Rochester (Other); Laval University (Other)
Responsible Party: Principal Investigator, Seth Lerner, Professor, Baylor College of Medicine
Other Study IDs: H-20395; 5P50CA091846 (NIH); NCT00831558 (obsolete NCT alias)
Record Dates: First submitted 2009-02-19; First posted 2009-02-20 (Estimated); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Bladder Cancer
Keywords: Bladder cancer; Smokers; Hematuria
MeSH Terms: conditions — Urinary Bladder Neoplasms; Hematuria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Males: 60 years of age or older Smokers or history of smoking
  Interventions: Other: Specimen and questionnaires only

INTERVENTIONS:
Other: Specimen and questionnaires only — Specimen and questionnaires only

SUMMARY:
In the study proposed, up to 1,500 men age 60 and over with strong smoking histories will test their urine for the presence of blood daily for two 10-day testing periods with the Ames Hemastix. Individuals with even a solitary positive test will undergo a thorough urologic evaluation to determine the cause of hematuria and follow-up will continue for 2 years after completion of the study.

DETAILED DESCRIPTION:
Reduction of cancer mortality is a stated goal of the National Cancer Institute. Cancer of the bladder is the 4th most commonly diagnosed cancer and 7th leading cause of cancer death in the American men, and represents an important target for mortality-reducing efforts. Furthermore, these tumors, even in early (i.e. curable) stages, usually cause several easily detectable abnormalities, including hematuria, and the presence of abnormal tumor products that are shed into urine or lie within exfoliated malignant cells.

The overall goal of the proposed study is to gain information concerning the performance characteristics of three bladder cancer markers when combined with hematuria testing in detecting bladder cancer.

A mail back questionnaire, completed at the beginning of the study, will provide information about the participants and the results of testings will be reported after each testing period. Individuals with even a solitary positive test will undergo a thorough urologic evaluation to determine the cause of hematuria and follow-up will continue or 2 years after completion of the study. At the time of the evaluation, three bladder cancer marker tests, NMP22 Bladder Chek, ImmunoCyt and UroVysion FISH will be performed, but regardless of the results, a hematuria evaluation will be completed. Data will be updated continually.

The 10 day testing with Hemastix will be repeated 9 months after the first one is completed regardless of the outcome of the first testing.

ELIGIBILITY:
Inclusion Criteria:

* Men age 60 and over, - who are current cigarette smokers OR - who have a history of at least 20 pack years smoking OR - who have over a 30 pack/year history who have stopped smoking within 10 years of the registration date OR - who have a 40 pack year history of smoking regardless of the quit date, will be eligible for participation.
* Patients with prostate or renal cancer must have been treated more than 5 years previously and be considered disease-free at the time of entry. In the case of prostate cancer, patients may have only received prostatectomy as their treatment and must have undetectable PSA's at study entry.
* In the case of calculus disease, patients must be believed to be stone free at time of study entry and could not have had a stone attack within the previous 2 years.
* Patients receiving anticoagulation therapy, such as Warfarin, Plavix, Lovenox, aspirin, etc. will be able to take part in the study and, will be thoroughly worked-up if the only explainable cause of hematuria is receiving anticoagulation medication.

Exclusion Criteria:

* history of urothelial cancer
* any malignancy other than non-melanoma skin cancers treated within the past 5 years
* benign tumors of the urinary tract that are still existent
* known urinary calculi
* medical or oncological conditions known to produce hematuria (e.g. glomerulonephritis, treatments with cyclophosphamide, methotrexate and pelvic radiation therapy)
* visual, psychological, neurological, musculoskeletal, etc. impairments that would make home testing impractical

Min Age: 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MD Anderson Cancer Center, Baylor College of Medicine, University of Rochester Medical Center and Laval University that contain within them county hospitals, Veterans Administrations Hospitals, fee-for-service clinics, and tertiary care facilities will enroll subjects. Each site will devise their own means of soliciting participants in the study.
Sampling Method: Probability Sample
Enrollment: 197 (Actual)
Dates: Start 2007-03; Primary Completion 2012-01 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Since the marker tests will only be administered to individuals with a positive Hemastix test, these are eight possible outcomes (one case with all negative marker tests and seven cases with as least one positive marker tests). | After last subject completes the study.

CONTACTS AND LOCATIONS:
Overall Officials: Seth P. Lerner, MD, Principal Investigator — Baylor College of Medicine
Locations (3):
- United States (2):
  - University of Rochester Medical Center, Rochester, New York
  - M.D. Anderson Cancer Center, Houston, Texas
- Laval University, Québec, Quebec, Canada